CLINICAL TRIAL: NCT03233789
Title: Entwicklung Und Validierung Eines ADL-Scores (Activities of Daily Life) Auf Basis Von FIM (Functional Independence Measure) Und EBI (Erweiterter Barthel-Index)
Brief Title: Development and Validation of an ADL-score Based on FIM and EBI
Acronym: EVA
Status: Completed | Type: Observational
Sponsor: Martin Brünger (Other)
Collaborators: Association nationale pour le développement de la qualité dans les hôpitaux et les cliniques (ANQ), Bern, Switzerland (Unknown)
Responsible Party: Sponsor-Investigator, Martin Brünger, Investigator, Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Other Study IDs: ANQ-FIM-EBI; U1111-1223-6650 (Other: World Health Organization)
Record Dates: First submitted 2017-07-25; First posted 2017-07-31 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Neurologic Disorder; ICF; Medical Rehabilitation; Assessment; Functional Independence; Observational Study
MeSH Terms: conditions — Nervous System Diseases | interventions — Neurological Rehabilitation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: neurologic rehabilitation — in-patient rehabilitation of neurologic disorders

SUMMARY:
The aim of this mixed-methods-study is to develop and validate an algorithm to transform FIM (Functional Independence Measure) and EBI (Extended Barthel Index) into an ADL score (Activities of Daily Life) that can be used to compare outcome quality of rehabilitation clinics.

The following steps are performed:

1. Development of an ADL-algorithms by experts
2. Validation of the ADL-algorithms in a quantitative approach
3. Finalization of the ADL-algorithms by experts based on study results

ELIGIBILITY:
Inclusion Criteria:

* Admission to in-patient neurologic rehabilitation clinic

Exclusion Criteria:

* No sufficient language skills (German, French or Italian)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with neurologic disorders in in-patient rehabilitation
Sampling Method: Probability Sample
Enrollment: 265 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2017-02-24 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Agreement FIM-based ADL-score vs. EBI-based ADL-score | within 3 days of admission to rehabilitation clinic
  Agreement according to Cohens kappa (FIM-based ADL-score vs. EBI-based ADL-score)

SECONDARY OUTCOMES:
Correlation FIM-based ADL-score vs. EBI-based ADL-score | within 3 days of admission to rehabilitation clinic
  Spearman's correlation (FIM-based ADL-score vs. EBI-based ADL-score)
Difference in FIM-based ADL-score vs. EBI-based ADL-score | within 3 days of admission to rehabilitation clinic
  Delta in points FIM-based ADL-score vs. EBI-based ADL-score

CONTACTS AND LOCATIONS:
Overall Officials: Karla Spyra, Prof. Dr., Study Director — Charite University, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No